CLINICAL TRIAL: NCT02914704
Title: Treatment of Benign Uterine Disorders Using High Intensity Focused Ultrasound (MR-HIFU)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN-HIFU
Record Dates: First submitted 2016-01-05; First posted 2016-09-26 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Uterine Fibroids; Adenomyosis
MeSH Terms: conditions — Leiomyoma; Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (1):
- Patients treated with MRI-HIFU (Experimental)
  Interventions: Device: MRI-HIFU

INTERVENTIONS:
Device: MRI-HIFU — Treatment of uterine fibroids with MRI-HIFU

SUMMARY:
MRI-guided high intensity focused ultrasound (MRI-HIFU) has been proven to be a safe and effective method in treating uterine fibroids and also adenomyosis. However, systematic studies on the effect of this treatment on factors affecting fertility are still lacking. Also quite little is known about body's systemic response to MRI-HIFU. Thus the aim of this study is to obtain more information on the systemic response of the body to the HIFU-treatment when treating non-malignant disease as well as to study the effect of MRI-HIFU on factors affecting fertility. Women with symptomatic uterine fibroids or adenomyosis suitable for MRI-HIFU treatment are recruited to this study. The severity of symptoms will be assessed with UFS-QoL and the same questionnaire will also be used in follow-up 3, 6 and 12 months after treatment. Blood, urine and endometrium samples will be collected pre- and postoperatively and during follow-up 3, 6 and 12 months after the treatment. From these samples detailed analysis of the immunological, inflammatory and hormonal response will be performed. As this is the first study in Finland of treating uterine fibroids and adenomyosis using MRI-HIFU, also a report about the efficacy of the MRI-HIFU in treating the uterine disorders will be published, and a key tool in assessing the treatment outcome would be the UFS-QoL questionnaire.

Also new methods for improving patient selection as well as treatment efficacy will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35
* Premenopausal
* Uterine size <20 gw
* Willingness to participate to the research
* Uterine fibroids with typical symptoms
* Maximum of 4 treated fibroids
* Dominant fibroid >2.5cm
* >50% of the fibroid is treatable

Exclusion criteria

* Unspecified pelvic tumours or ovarian masses, PID
* Major corrective surgery to uterus (simple myomectomy excluded)
* Major uterine anomalies
* Unability to calculate the volume of uterine fibroids
* Marked uterine calcification
* Marked scarring of the lower abdomen
* Suspicion of malignancy
* Marked general health problem contraindicating MRI
* Claustrophobia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Technical efficacy of HIFU for treatment of uterine fibroids as assessed by a change in the Symptom Severity Score | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi M Joronen, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided